CLINICAL TRIAL: NCT02899507
Title: Prophylactic Versus Clinically-driven Antibiotics in Comatose Survivors of Out-of-hospital Cardiac Arrest
Brief Title: Prophylactic Antibiotics in Comatose Survivors of Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Marko Noc, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P3-0331
Record Dates: First submitted 2016-06-30; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-08

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Out-of-hospital cardiac arrest; Prophylactic antibiotics
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic antibiotic (Experimental): Amoxicillin-Clavulanic acid 1.2g every 8h
  Interventions: Drug: Amoxicillin-Clavulanic acid
- Clinically-driven antibiotics (No Intervention): Administration of antibiotics in clinically-driven group was at the discretion of attending intensivist. Selection of antibiotic in clinically-driven group was empirical or based on the results of bacterial cultures if already available.

INTERVENTIONS:
Drug: Amoxicillin-Clavulanic acid — Patients without evidence of tracheobronchial aspiration were randomized to immediate prophylactic Amoxicillin-Clavulanic acid 1,2 gr/8h
  Other Names: Amoksiklav, Augmentin
  Arms: Prophylactic antibiotic

SUMMARY:
The purpose of this study is to determine whether there is potential benefits of prophylactic antibiotic treatment in comatose survivors of out-of-hospital cardiac arrest (OHCA) treated in intensive care unit with therapeutic hypothermia.

DETAILED DESCRIPTION:
Postresuscitation management of comatose survivors of out-of-hospital cardiac arrest (OHCA) significantly improved and "bundle of care" including therapeutic hypothermia, immediate coronary angiography, percutaneous coronary intervention (PCI) and contemporary intensive care nowadays leads to survival with good neurological recovery. Benefit of prophylactic antibiotics, which may suppress development of postresuscitation infection and especially early onset pneumonia and thereby decrease the severity of postresuscitation systemic inflammatory response, is controversial. Because of these uncertainties, the investigators performed a single-center randomized clinical trial comparing prophylactic versus clinically-driven administration of antibiotics in comatose survivors of OHCA. The investigators hypothesized that prophylactic antibiotics may decrease the severity of postresuscitation systemic inflammatory response by reducing the incidence of postresuscitation infection and especially pneumonia which was further addressed by repeat microbiological sampling.

ELIGIBILITY:
Inclusion Criteria:

* Female and male over 18 years old
* Comatose survivors of out-of-hospital cardiac arrest treated in intensive care unit with therapeutic hypothermia

Exclusion Criteria:

* Suspected or confirmed pregnancy
* Allergy to amoxicillin-clavulanic acid
* Tracheobronchial aspiration
* Antibiotic therapy before cardiac arrest
* Need of antibiotics due to other causes
* Candidates for immediate veno-arterial extracorporeal membrane oxygenation (VA ECMO)
* Patients in whom no active treatment was decided on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Value of C-reactive protein (CRP) at day three | Three days after admission to Intensive care unit (ICU)
  Expressed in milligram/litre (normal <5 mg/L)

SECONDARY OUTCOMES:
Severity of systemic inflammatory response estimated by peak white blood cell count (WBC) | First measurement at admission in hospital and afterwards in 24 hours intervals during stay in the intensive care unite (ICU) but not longer then first seven days
  Expressed in number of white blood cells x 109 per litre (L)
Severity of systemic inflammatory response estimated by peak value of procalcitonin (PCT) | First measurement at admission in hospital and afterwards in 24 hours intervals during stay in the intensive care unite (ICU) but not longer then first seven days
  Expressed in microgram/litre (normal <0.5 microgram/L)
Severity of systemic inflammatory response estimated by peak value of neutrophil Cluster of differentiation 64 (CD 64) | First measurement at admission in hospital and afterwards in 24 hours intervals in the first three days
  Neutrophil CD 64 expression was used as an index of sepsis with >1.2 indicating greater likelihood of sepsis
Appearance of pneumonia on chest X ray | Chest X ray was taken on admission and afterwards on daily basis during the stay in the intensive care unite but not longer than first week
Incidence of positive blind mini bronchoalveolar lavage (Mini-BAL) on day 3 | Mini-BAL was performed on the third day after the sudden cardiac arrest
Incidence of positive hemocultures | From the admission until the patient was transferred to the ward. This was always during the ICU stay-one month
Duration of tracheal intubation | From the day of admission until the extubation. This was always during the ICU stay- one month
  Duration of intubation was expressed as days of intubation started with admission until the extubation. Because this is being done in intensive care unite, the time frame is duration of ICU stay
Duration of mechanical ventilation | From the admission until spontaneous breathing . This was during ICU stay-one month
  Duration of mechanical ventilation was expressed as days the patient needed the mechanical support for breathing regardless of mode of support
ICU stay | From the admission until the patient was transferred to ward, usually less than one month
Survival with good neurological outcome | Up to six months after the event
  Good neurological outcome was characterised using cerebral performance category (CPC) with 1-2 indicating good neurological recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Noč, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomte O, Andersen GO, Jacobsen D, Draegni T, Auestad B, Sunde K. Strong and weak aspects of an established post-resuscitation treatment protocol-A five-year observational study. Resuscitation. 2011 Sep;82(9):1186-93. doi: 10.1016/j.resuscitation.2011.05.003. Epub 2011 May 14. PMID 21636202
- [Background] Stub D, Hengel C, Chan W, Jackson D, Sanders K, Dart AM, Hilton A, Pellegrino V, Shaw JA, Duffy SJ, Bernard S, Kaye DM. Usefulness of cooling and coronary catheterization to improve survival in out-of-hospital cardiac arrest. Am J Cardiol. 2011 Feb 15;107(4):522-7. doi: 10.1016/j.amjcard.2010.10.011. Epub 2010 Dec 22. PMID 21184989
- [Background] Kocjancic ST, Jazbec A, Noc M. Impact of intensified postresuscitation treatment on outcome of comatose survivors of out-of-hospital cardiac arrest according to initial rhythm. Resuscitation. 2014 Oct;85(10):1364-9. doi: 10.1016/j.resuscitation.2014.06.028. Epub 2014 Jul 8. PMID 25010782
- [Background] Perbet S, Mongardon N, Dumas F, Bruel C, Lemiale V, Mourvillier B, Carli P, Varenne O, Mira JP, Wolff M, Cariou A. Early-onset pneumonia after cardiac arrest: characteristics, risk factors and influence on prognosis. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1048-54. doi: 10.1164/rccm.201102-0331OC. PMID 21816940
- [Background] Mongardon N, Perbet S, Lemiale V, Dumas F, Poupet H, Charpentier J, Pene F, Chiche JD, Mira JP, Cariou A. Infectious complications in out-of-hospital cardiac arrest patients in the therapeutic hypothermia era. Crit Care Med. 2011 Jun;39(6):1359-64. doi: 10.1097/CCM.0b013e3182120b56. PMID 21336107
- [Background] Gajic O, Festic E, Afessa B. Infectious complications in survivors of cardiac arrest admitted to the medical intensive care unit. Resuscitation. 2004 Jan;60(1):65-9. doi: 10.1016/j.resuscitation.2003.08.005. PMID 14987786
- [Background] Woo JH, Lim YS, Yang HJ, Park WB, Cho JS, Kim JJ, Hyun SY, Lee G. Factors associated with pneumonia in post-cardiac arrest patients receiving therapeutic hypothermia. Am J Emerg Med. 2014 Feb;32(2):150-5. doi: 10.1016/j.ajem.2013.10.035. Epub 2013 Oct 26. PMID 24268585
- [Derived] Ribaric SF, Turel M, Knafelj R, Gorjup V, Stanic R, Gradisek P, Cerovic O, Mirkovic T, Noc M. Prophylactic versus clinically-driven antibiotics in comatose survivors of out-of-hospital cardiac arrest-A randomized pilot study. Resuscitation. 2017 Feb;111:103-109. doi: 10.1016/j.resuscitation.2016.11.025. Epub 2016 Dec 14. PMID 27987397